CLINICAL TRIAL: NCT02890485
Title: The Effects of Dry Needling on Patients with Knee Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Matt Briggs, Assistant Professor-Practice, Ohio State University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016H0003
Record Dates: First submitted 2016-08-29; First posted 2016-09-07 (Estimated); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Patellofemoral Pain Syndrome; Anterior Knee Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Dry Needling; Physical Therapy Modalities; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Glute Dry Needling (Experimental): Receives dry needling to their gluteal muscles in addition to standard physical therapy treatment.
  Interventions: Device: Dry Needling
- Quad Dry Needling (Experimental): Receives dry needling to their quadriceps muscles in addition to standard physical therapy treatment.
  Interventions: Device: Dry Needling
- Glute Sham Dry Needling (Sham Comparator): Receives sham dry needling to their gluteal muscles in addition to standard physical therapy treatment.
  Interventions: Device: Sham Dry Needling
- Quad Sham Dry Needling (Sham Comparator): Receives sham dry needling to their quadriceps muscles in addition to standard physical therapy treatment.
  Interventions: Device: Sham Dry Needling
- Control (Active Comparator): Receives only standard physical therapy treatment.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Device: Dry Needling — Dry needling consists of small, monofilament needles that are administered directly into the tissue and manipulated to make the muscle relax for pain relief. This technique is used to treat dysfunctions in skeletal muscle and connective tissue to help diminish pain, reduce impairments of body structure and restore function. Dry needling will be performed in the gluteal or the quadriceps muscle groups depending upon group randomization.
  Other Names: Trigger Point Acupunture
  Arms: Glute Dry Needling; Quad Dry Needling
Device: Sham Dry Needling — The same overall procedures will be used as in the "true" dry needling groups and applied to the same muscle groups (gluteal or quadriceps) depending upon ground randomization. Sham dry needling will be performed using a commercially available sham needling system commonly.This set-up utilizes a blunt tipped needle. When the sham needle is pressed downward, the barrel of the needle retracts into the handle, giving the appearance of insertion of the needle through the skin. This also creates pressure on the subject's skin, increasing the sensation of dry needling. Patients will not be allowed to observe the areas being needled or sham needled.
  Arms: Glute Sham Dry Needling; Quad Sham Dry Needling
Other: Physical Therapy — Physical Therapy and exercise as determined by the examining clinician based on the patients specific impairments and functional limitations. All subjects enrolled in this study will receive an initial physical therapy (PT) evaluation and then 2 additional PT sessions a week a part. Interventions and prescribed home exercises will be specific to the patients' primary individual impairments as determined during the initial PT evaluation. These interventions reflect current evidence, but will not be restrictive to specific exercises; prescribed exercises will be deemed appropriate based on the treating PTs' examination, evaluation, and identification of each patients' primary deficits, impairments, functional limitations, and current literature.
  Other Names: Exercise
  Arms: Control

SUMMARY:
This study is testing the effectiveness of "dry needling" for pain management and on muscle strength and leg function for those with knee pain. Dry needling consists of small, monofilament needles that are administered directly into the tissue and manipulated to make the muscle relax for pain relief. This technique is used to treat dysfunctions in skeletal muscle and connective tissue to help diminish pain, reduce impairments of body structure and restore function.

DETAILED DESCRIPTION:
This project will evaluate the effects of dry needling on pain, muscle performance, and function in those with patellofemoral pain syndrome (PFPS) of the knee. Variables of interest will include self-reported pain scores, self-reported functional outcome and disability questionnaire scores, and various objective clinical measures including muscle strength, joint range of motion, and movement patterns during basic tasks related to activities of daily living. Patients who are referred to physical therapy with PFPS will be recruited. Patients will be randomly and equally allocated into one of the following groups: 1. Gluteal dry needling (GLUTE) 2. Quadriceps dry needling (QUAD) 3. Sham gluteal dry needling (SHAM GLUTE) 4. Sham quadriceps dry needling (SHAM QUAD) 5. Control group (CONTROL) Groups 1-4 will receive 2 sessions of dry needling or sham dry needling to the gluteal and/or quadricpes muscles on their painful lower limb over 2 consecutive weeks in addition to standard physical therapy. The CONTROL group will only receive standard physical therapy. The sham treatment groups (groups 3-4) will receive a placebo treatment that does not penetrate the skin or muscles. Measurements will be performed at baseline prior to any physical therapy interventions and then at week 3.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years-of-age
* Referred for physical therapy
* Presence of anterior knee pain around the patella during ascending/descending stairs, squatting, and/or running for at least 3 months.

Exclusion Criteria:

* Unable to provide consent
* Bilateral patellofemoral pain syndrome
* Received previous dry needling treatments
* Pregnancy
* History of pain less than 3 months
* Imaging demonstrating the presence of confounding internal abnormality (e.g. chondral defects, ligamentous injury, and/or meniscal pathology),
* Patellar instability
* Presence of a neurological condition that would affect movement
* Contraindications to dry needling techniques (e.g. a history of bleeding disorders, phobia of needles, an active cancer diagnosis, and presence of other systemic illness such as fever or signs of infection)
* Actively receiving treatment for knee pain outside of the current study protocol while enrolled in the study;
* received active and supervised PT treatment for knee pain within the last 4 weeks;
* history of knee surgery less than 6 months ago
* history of surgical correction of the patellofemoral complex (e.g. MPFL reconstruction, patellar realignment surgery, etc)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-08; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Anterior Knee Pain Scale (AKPS) score to 3 weeks | Baseline and Post testing (week 3)
  The AKPS is commonly used to evaluate function in patients with PFPS. It is a 13-item questionnaire with a maximum score of 100. Higher scores are indicative of better function. The minimal detectable change (MDC) and the minimal clinically important difference (MCID) of the AKPS has been reported to be 10 and 13 points respectively and has high test-retest reliability (ICC: 0.81 to 0.95). The standard error of measurement is 3 and has been shown to be valid (0.92).
Change from Baseline Numeric Pain Rating Scale (NPRS) score to 3 weeks | Baseline and Post testing (week 3)
  Pain will be measured using the numeric pain rating scale (NPRS). Patients will be asked to rate their pain on 11-point (0-10) scale with 0 being no pain and 10 being extreme pain. The NPRS is a common measure of pain in patients with PFPS and has been shown to be reliable and responsive (minimal clinically important difference = 2 points).

SECONDARY OUTCOMES:
Change from Baseline Lateral step-down (LSD) test score to 3 weeks | Baseline and Post testing (week 3)
  the LSD test will also be performed to evaluate movement quality. Two-dimensional video analysis and scoring will be conducted during the LSD test. Participants will be asked to stand with their stance foot close to the edge of a 20cm step and place their second toe over a white piece of tape, while their non-stance limb is off the side of the step. Participants will be asked to keep both hands on their waist and bend their knee until the heel of their uninvolved leg lightly touched the floor, then to immediately return to the starting position. Participants will be instructed to perform 5 trials and will be scored on the 4th trial. Immediately following the test, participants will rate any knee pain experienced during the test as described above. The LSD test has been shown to have moderate reliability.
Change from Baseline Isometric knee and hip peak torque values to 3 weeks | Baseline and Post testing (week 3)
  Isometric knee and hip peak torque will be measured for knee extension, knee flexion, hip abduction, and hip extension using a Biodex System III dynamometer (Biodex Medical Systems, Inc. Shirley, New York, USA) on each subject's pain and non-painful limb . A standardize set-up and protocol commonly performed in clinical care and based on manufacture guidelines will be used. Peak torque during each task will be recorded as absolute values (Nm) and normalized to body mass (Nm/kg). The data from the strength testing will be used to power future studies evaluating the effects of dry needling on muscle force generation.
Change from Baseline Lower Extremity Functional Scale (LEFS) score to 3 weeks | Baseline and Post testing (week 3)
  The LEFS is commonly used self report questionnaire to evaluate function in patients with patellofemoral pain syndrome (PFPS) and other lower extremity problems.
Change from Baseline Pressure Pain Threshold to 3 weeks | Baseline and Post testing (week 3)
  Pressure pain threshold (PPT) will be used to measure pain sensitivity and potential abnormalities in pain processing. PPT measures have been shown to have excellent intra-rater (ICC=0.94-0.97) and inter-rater reliability (ICC=0.72-0.90). A digital pressure algometer will be used to measure PPT at 5 sites [3 sites around the patella, 1 site at the center of the patella, and 1 site on the tibialis anterior].

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S Briggs, DPT, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No